CLINICAL TRIAL: NCT01486524
Title: A Multicenter Pharmacogenomic Biomarker Study in Matched Patients With Severe Sepsis Treated With or Without Recombinant Human Activated Protein C [Xigris®, Drotrecogin Alfa (Activated)]
Brief Title: Pharmacogenomic Biomarker Study for Recombinant Human Activated Protein C Treatment in Severe Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sirius Genomics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SGX301
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: pharmacogenomic biomarker; predictive marker; prospective-retrospective; propensity score; matched-patients trial
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Minimum 700 ng DNA required, extracted from blood samples. Two Improved Response Polymorphisms (IRPs) will be tested in this study. IRP A is comprised of two single nucleotide polymorphisms (SNPs), RYR2 (ryanodine receptor 2 gene) rs684923 and ACIN1 (apoptotic chromatin condensation inducer 1 gene)rs3751501. IRP B is comprised of two SNPs, SPATA7 (spermatogenesis associated 7 gene) rs3179969 and FLI1 (Friend leukemia virus integration 1 gene) rs640098. An individual patient will be considered to be biomarker positive if they have the responsive genotype for either of the SNPs or for both of the SNPs in the IRP.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DrotAA Treatment Group: Patients with severe sepsis at high risk of death (INDICATED patients) who received treatment with drotrecogin alfa (activated (DrotAA) as part of standard care in ICU. The standard dosing regimen for DrotAA is 96 hours of continuous infusion at a dose of 24 ug/kg/hour. DrotAA is also known as recombinant human activated protein C.
- Control Group (non-DrotAA treated): Patients with severe sepsis at high risk of death (INDICATED patients) who did not receive DrotAA treatment as part of their standard care in an ICU. The Control group patients will be selected to match the DrotAA-treated patients based on numerous clinical covariates, including propensity score (for DrotAA treatment).

SUMMARY:
The overall purpose of the study is to determine whether either of the Improved Response Polymorphisms (IRPs) individually predicts a differential DrotAA treatment effect in patients with severe sepsis and high risk of death. This will be an international, multicenter, "prospective-retrospective", nonrandomized, controlled, outcome-blinded, genotype-blinded, matched-patients study. No prospective enrollment or treatment of patients will occur under this protocol. Retrospectively collected clinical data and DNA samples will be analyzed for existing cohorts of patients with severe sepsis who were previously treated with DrotAA (treatment group) or not (control group) as part of their standard care in an ICU.

DETAILED DESCRIPTION:
This will be a multicenter, "prospective-retrospective", controlled, matched-patients study. Retrospective phenotypic data and DNA samples will be obtained from patient registries and clinical trials where the study hypotheses were not related to DrotAA treatment. The prospective aspect of this study will be the statistical testing of prespecified hypotheses regarding the IRP genotype as a predictive biomarker for differential DrotAA treatment effects.

To control for differences in standard of care in different countries and medical centers, the selection of matched control patients will be performed within each cohort. Control patients will be selected to match the DrotAA-treated patients using an algorithm that matches on baseline demographic and disease characteristics that may have influenced the decision to give DrotAA or that may impact survival. A propensity score (the likelihood for having received DrotAA treatment) will be derived using the matching variables that are common in all cohorts. The number of matched control patients for each treated patient will be variable, up to a maximum of 3.

The selection of the control patients via the matching algorithm will be conducted by an independent clinical research organization (CRO) in a blinded manner - specifically without knowledge of survival outcome, other outcome data, and genotype. A two-phase transfer of data from each center will be implemented to ensure that the selection of matched control patients is implemented in a blinded manner. The first step will involve the transfer of the baseline data for all variables needed to conduct the matching. Once the control patients have been identified for each cohort, the outcomes data will be transferred to the CRO in the second phase of data transfer.

Centralized genotyping using a validated Taqman®-based analytical method will be conducted on the DNA samples for all matched patients. The genotyping laboratory will be blinded to treatment and outcome.

The total number of patients in the available cohorts is >23,000, with approximately 800 who have received DrotAA as part of their standard ICU-based care. After applying eligibility criteria to all patients and selecting the matched control patients, it is expected that the final analysis will include approximately 3000 patients.

ELIGIBILITY:
Inclusion Criteria for INDICATED population:

1. Age ≥ 18 years
2. Severe sepsis (must meet a, b, and c below)

   * Suspected or proven infection
   * Systemic Inflammatory Response Syndrome (SIRS)(must meet 2 of 4 criteria)

     * Temperature < 36°C or > 38°C
     * Heart rate > 90 beats/minute
     * Respiratory rate > 20 breaths/minute or PaC02 < 32 mm Hg) or on mechanical ventilation
     * White blood cell count < 4,000/mm3 or > 12,000/mm3
   * At least one organ dysfunction due to sepsis based on definitions of clinically significant organ dysfunction

     * Cardiovascular dysfunction [must meet one of (1), (2), or (3) below]:

       * Systolic blood pressure ≤ 90 mmHg and pH ≤ 7.3
       * Mean arterial pressure ≤ 70 mmHg and pH ≤ 7.3
       * Reported use of a vasopressor alone is sufficient evidence of shock
     * Pulmonary dysfunction: PaO2/FiO2 ≤ 300 mmHg
     * Central Nervous System dysfunction: Glasgow Coma Scale ≤ 12
     * Coagulation dysfunction: platelets ≤ 80,000/mm3
     * Renal dysfunction: creatinine ≥ 2.0 mg/dL
     * Hepatic dysfunction: bilirubin ≥ 2.0 mg/dL
3. High risk of death (one of a, b, or c below)

   * APACHE II ≥ 25
   * SAPS II ≥ 54
   * Multiple organ dysfunction - two or more clinically significant organ dysfunctions (as defined above), which have occurred within 2 days of each other
4. Platelet counts ≥ 30,000/mm3
5. DrotAA status known

Exclusion Criteria:

1. Patients with no DNA
2. Patients enrolled in local cohort more than 2 years before Xigris [drotrecogin alfa activated)] was commercially available

A secondary analysis population with severe sepsis will be defined by Inclusion Criteria 1, 2, 4, and 5 above, and the Exclusion Criteria. This will be referred to as the SEVSEP population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The indicated-patients population (INDICATED) population will be the primary population for this study and it will include those DrotAA-treated patients who have documented severe sepsis and high risk of death, defined in keeping with the regulatory approvals in the EU and US, and their matched controls. Documented organ dysfunction will be defined according to published criteria. A secondary severe sepsis population (SEVSEP) will have had documented severe sepsis, but not necessarily a high risk of death. The INDICATED population will be a subset within the broader SEVSEP population.The SEVSEP population will be analyzed only if at least 10% larger than the INDICATED population.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality through Day 28 | Through Day 28.
  All cause in-hospital mortality up to Day 28 or discharge, whichever comes first. Day 1 is the day when patient meets eligibility criteria for this study.

SECONDARY OUTCOMES:
Time to death in hospital | Through Day 28
  Time to death (any cause) in hospital, censored by the competing risk of discharge from hospital
Time to death | Through Day 60
  Time to death (any cause), censored at Day 60 or last evaluation. Will be evaluated using data from centers where follow-up extended beyond hospital discharge.
Mechanical ventilator-free days through Day 28 | Through Day 28
  Number of days alive and free of mechanical ventilation from Day 1 through Day 28.
ICU-free days through Day 28 | Through Day 28
  Number of days alive and free of ICU from Day 1 through Day 28.
Hospital-free days through Day 28 | Through Day 28
  Number of days alive and free of hospitalization from Day 1 through Day 28.
ICU length of stay | Through Day 180
Hospital length of stay | Through Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD, PhD, Principal Investigator — University of Versailles; Alexandra DJ Mancini, MSc, Study Director — Sirius Genomics Inc.
Locations (8):
- United States (4):
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Bayview Medical Center, Baltimore, Maryland
  - Harvard University School of Public Health, Boston, Massachusetts
  - Vanderbilt University Schoo of Medicine, Nashville, Tennessee
- University of British Columbia and Providence Health Care, St. Paul's Hospital, Vancouver, British Columbia, Canada
- France (2):
  - University of Versailles, Hospital Raymond Poincaré (AP-HP), Garches
  - Université Paris Descartes, Sorbonne Paris Cité, Cochin Hotel-Dieu University Hospital, Paris
- Imperial College London, Charing Cross Hospital, London, United Kingdom

REFERENCES:
- [Derived] Annane D, Mira JP, Ware LB, Gordon AC, Hinds CJ, Christiani DC, Sevransky J, Barnes K, Buchman TG, Heagerty PJ, Balshaw R, Lesnikova N, de Nobrega K, Wellman HF, Neira M, Mancini ADJ, Walley KR, Russell JA. Pharmacogenomic biomarkers do not predict response to drotrecogin alfa in patients with severe sepsis. Ann Intensive Care. 2018 Jan 31;8(1):16. doi: 10.1186/s13613-018-0353-2. PMID 29388048